CLINICAL TRIAL: NCT06088082
Title: "Analgesic Efficacy of Combined Transversus Abdominis Plane Block and Posterior Rectus Sheath Block in Patients Undergoing Laparoscopic Appendectomy"
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Saud Medical City (Other Government)
Responsible Party: Principal Investigator, Rashid Saeed Khokhar, consultant anesthetist, King Saud Medical City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: E-21-6173
Record Dates: First submitted 2023-05-16; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: ERAS
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: To evaluate the combined efficacy US-guided TAP block and PRS block in patients undergoing laparoscopic appendectomy.
  Early mobilization, opioid consumption, Postoperative Nausea & Vomiting (PONV), length of hospital stay (LOS), patient satisfaction in patients scheduled for laparoscopic appendectomy.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: . All patients, care providers in PACU & ward (nurses), and outcome assessors (assistant anesthesiologist) will be blinded to the group allocation. Only the assigned anesthesiologist responsible for perioperative care will be aware of the group allocation to treat any unwanted side effects during and after the
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTROL GROUP (No Intervention): ) will receive standard routine postoperative analgesia at our institute.
- TREATMENT GROUP (Experimental): The patients will be divided into two groups; group-1 (n= 50) will receive pre-procedure right US-guided TAP and bilateral PRS blocks with bupivacaine 0.25% 20 ml for TAP block and 10 ml for PRS block .
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — Patients will be randomly assigned to receive a TAP and PRS blocks with 34 mL of 0.25% bupivacaine (study group) or standard hospital analgesia protocol (control group).
  Other Names: TRASVERSE ABDOMINIS AND POSTERIOR RECTUS SHEATH BLOCKS
  Arms: TREATMENT GROUP

SUMMARY:
laparoscopic appendectomy is most common surgical procedure necessitates evidence-based clinical pathways such as Enhanced Recovery After Surgery (ERAS). The paradigm of surgery has been shifted from open to laparoscopic. Laparoscopic appendectomy is the most common procedure performed in our institute for acute and chronic appendicitis. Pain control in ERAS is one of the key factors for improved outcomes. Surgery induced acute postoperative pain, stress response, and fatigue lead to prolonged convalescence and hospital stay. Optimal titrated safe postoperative pain management in laparoscopic appendectomy patients remains a challenge.

DETAILED DESCRIPTION:
Objectives: To evaluate the efficacy of combined transversus abdominis plane (TAP) and posterior rectus sheath (PRS) blocks on perioperative pain, early mobilization, opioid consumption, Postoperative Nausea & Vomiting (PONV), length of hospital stay (LOS), patient satisfaction in patients scheduled for laparoscopic appendectomy Methods: 100 patients scheduled for Laparoscopic appendectomy will be recruited in this prospective randomized, blinded clinical study. The patients will be divided into two groups; group-1 (TAP and PRS blocks) (n= 50) will receive intraoperative combined TAP and PRS blocks with bupivacaine 0.25% 2-3 mg/kg, and Group 2 (standard care) (n= 50) will receive standard analgesic protocol in our institute. Intraoperatively, all patients will receive conventional intravenous (IV) analgesics and antiemetics (Paracetamol 1 gram + Lornoxicam 8 mg + Dexamethasone 8mg + Ondansetron 4mg). For breakthrough pain in Post Anesthesia Care Unit (PACU) and ward, all patients will be prescribed for IV PRN (as needed) morphine 2 mg maximum 10 mg, paracetamol 1 gram every 6 hours, lornoxicam 8 mg every 8 hours. During pre-anesthesia assessment patients will be instructed how to use 10 cm numerical rating scale (NRS) (0 cm no pain, 10 cm worse pain) to report pain postoperatively. On arrival to the operation room (OR), all eligible participants will have intravenous (IV) cannula in situ and monitors, according to the Association of Anesthetists of Great Britain and Ireland (AAGBI). Anesthesia will be induced with the following drugs: fentanyl 2mcg/kg, propofol 2mg/kg, followed by rocuronium 1mg/kg to facilitate tracheal intubation. Anesthesia drugs doses will be calculated according to ideal body weight (IBW) and adjusted body weight (AjBW) using this link: https://globalrph.com/medcalcs/adjusted-body-weight-ajbw-and-ideal-body-weight-ibw-calc/. General anesthesia will be maintained with Desflurane Minimum Alveolar Concentration (MAC) value of 0.7-1with Fraction of Inspired Oxygen (FIO2) 45%. Before skin incision, US guide left TAP and bilateral PRS blocks will be performed by the anesthesia consultant/senior registrar. and then at the end of surgical procedure desflurane will be discontinued and 2.5 mg of neostigmine with 0.4 micrograms of glycopyrolate will be given. All patients will be transferred to PACU after tracheal extubation. Patients will be monitored in PACU for hemodynamics, pain measured by NRS, morphine or any other analgesic consumption and for PONV antiemetics will be given as required. And in the ward 2, 6,12 and 24 hourly till discharged to home. Patients will be transferred to the ward from PACU when they achieve modified Aldrete score of 9 on two sequential measurements of 10 minutes' interval. All patients, care providers in PACU & ward (nurses), and outcome assessors (assistant anesthesiologist) will be blinded to the group allocation. Only the assigned anesthesiologist responsible for perioperative care will be aware of the group allocation to treat any unwanted side effects during and after the operation. And in the ward 2, 6,12 and 24 hourly pain score (NRS) will be assessed till discharged to home.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist [ASA] I-III patients
* Age 14-60 years
* Either gender
* Patients scheduled for laparoscopic appendectomy.
* Patient weight 50kg and above.

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status IV
* Patients with uncontrolled hypertension.
* Anticipated difficult intubation.
* Allergic to morphine
* Allergic to bupivacaine
* Clinically significant neurological, cardiovascular, renal hepatic disease planned for postoperative surgical intensive care (SICU) admission.
* History of drug abuse or chronic opioid use
* Laparoscopic procedure converted to open.
* The patient weighed 100 kg and above.
* Difficult anatomic landmarks on ultrasound scanning.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
to assess the pain score by verbal numerical rating scale[VNRS] | 7 months
  to assess the pain score by using verbal numerical rating scale [0-10]in immediate postop period on arrival in PACU and then after 2,4,6,12 and 24 hours postop.between two groups.Low scores on verbal numerical rating scale will be beneficial factor in early discharge of patients from the hospital.

SECONDARY OUTCOMES:
opiod consumption | 7 months
  to measure opiods consumption in milligrams[mg] during intraop followed in PACU and after 4,6,12 and 24 hours postop.
early mobility after surgery measured by john hopkins highest level of mobility scale[JH-HLM] | 7 months
  early mobility after surgery measured by john hopkins highest level of mobility scale[JH-HLM] this scale is a validated 1-item ordinal scale ranging from lying passively in bed[score=1] to walking equal or more than 250 feet [score=8] within immediate postop and within 24 hours postop.high scores on mobility scale used indicates early patient mobility and discharge from the hospital.
to assess the severity of postoperative [PONV] during immediate postop and after 4,6,12 and 24 hours postop. | 7 months
  to assess the severity of postoperative [PONV]
  during immediate postop and after 4,6,12 and 24 hours postop. by using numeral rating scale [0-10]for nausea as no for score 0,mild for 1-3,moderate for 4-6, and severe for 7-10 with propensity to vomiting.and document vomiting by yes or no.low scores on verbal numerical rating scale for nausea will be contributing early discharge of the patients from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: rashid khokhar, fcps, Principal Investigator — King Saud Medical City
Locations (1):
- Rashid Saeed Khokhar, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Robertson TC, Hall K, Bear S, Thompson KJ, Kuwada T, Gersin KS. Transversus abdominis block utilizing liposomal bupivacaine as a non-opioid analgesic for postoperative pain management. Surg Endosc. 2019 Aug;33(8):2657-2662. doi: 10.1007/s00464-018-6543-z. Epub 2018 Nov 2. PMID 30390161
- [Background] Moradkhani M, Hejri P, Nadri S, Beiranvand S. Effects of ADJUVANT Ketamine on Induction of Anesthesia for the Cesarean Section. Curr Rev Clin Exp Pharmacol. 2021;16(2):197-200. doi: 10.2174/1574884715666200310103317. PMID 32156239
- [Background] Alizadeh R, Aghsaie Fard Z. Renal impairment and analgesia: From effectiveness to adverse effects. J Cell Physiol. 2019 Aug;234(10):17205-17211. doi: 10.1002/jcp.28506. Epub 2019 Mar 27. PMID 30916404
- [Background] Beiranvand S, Karimi A, Vahabi S, Amin-Bidokhti A. Comparison of the Mean Minimum Dose of Bolus Oxytocin for Proper Uterine Contraction during Cesarean Section. Curr Clin Pharmacol. 2019;14(3):208-213. doi: 10.2174/1574884714666190524100214. PMID 31124424
- [Background] Ma N, Duncan JK, Scarfe AJ, Schuhmann S, Cameron AL. Clinical safety and effectiveness of transversus abdominis plane (TAP) block in post-operative analgesia: a systematic review and meta-analysis. J Anesth. 2017 Jun;31(3):432-452. doi: 10.1007/s00540-017-2323-5. Epub 2017 Mar 7. PMID 28271227
- [Background] Beiranvand S, Sorori MM. Pain management using nanotechnology approaches. Artif Cells Nanomed Biotechnol. 2019 Dec;47(1):462-468. doi: 10.1080/21691401.2018.1553885. PMID 30688094
- [Background] Tupper-Carey DA, Fathil SM, Tan YK, Kan YM, Cheong CY, Siddiqui FJ, Assam PN. A randomised controlled trial investigating the analgesic efficacy of transversus abdominis plane block for adult laparoscopic appendicectomy. Singapore Med J. 2017 Aug;58(8):481-487. doi: 10.11622/smedj.2016068. Epub 2016 Apr 8. PMID 27056207
- [Background] Alizadeh R, Mireskandari SM, Azarshahin M, Darabi ME, Padmehr R, Jafarzadeh A, Aghsaee-Fard Z. Oral clonidine premedication reduces nausea and vomiting in children after appendectomy. Iran J Pediatr. 2012 Sep;22(3):399-403. PMID 23400517
- [Background] Khoo CK, Vickery CJ, Forsyth N, Vinall NS, Eyre-Brook IA. A prospective randomized controlled trial of multimodal perioperative management protocol in patients undergoing elective colorectal resection for cancer. Ann Surg. 2007 Jun;245(6):867-72. doi: 10.1097/01.sla.0000259219.08209.36. PMID 17522511
- [Background] Muller S, Zalunardo MP, Hubner M, Clavien PA, Demartines N; Zurich Fast Track Study Group. A fast-track program reduces complications and length of hospital stay after open colonic surgery. Gastroenterology. 2009 Mar;136(3):842-7. doi: 10.1053/j.gastro.2008.10.030. Epub 2008 Nov 1. PMID 19135997
- [Background] Stokes AL, Adhikary SD, Quintili A, Puleo FJ, Choi CS, Hollenbeak CS, Messaris E. Liposomal Bupivacaine Use in Transversus Abdominis Plane Blocks Reduces Pain and Postoperative Intravenous Opioid Requirement After Colorectal Surgery. Dis Colon Rectum. 2017 Feb;60(2):170-177. doi: 10.1097/DCR.0000000000000747. PMID 28059913
- [Background] Beverly A, Kaye AD, Ljungqvist O, Urman RD. Essential Elements of Multimodal Analgesia in Enhanced Recovery After Surgery (ERAS) Guidelines. Anesthesiol Clin. 2017 Jun;35(2):e115-e143. doi: 10.1016/j.anclin.2017.01.018. PMID 28526156